CLINICAL TRIAL: NCT00012753
Title: Automated Calls With Nurse Follow-Up to Improve Diabetes Ambulatory Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 95-084
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Automated telephone health status assessments with nurse follow-up.

INTERVENTIONS:
Procedure: Automated telephone health status assessments with nurse follow-up.

SUMMARY:
Regular outpatient follow-up is important for all diabetes patients, with some needing frequent attention because their health is unstable, their treatment regimen is complex, or their social supports are inadequate. However, many patients live with access barriers that limit their use of outpatient services, fail to attend outpatient appointments, and experience worse outcomes than trials of aggressive management suggest is possible. Although labor-intensive, telephone care programs are one potential strategy for bringing diabetes management services into patients� homes and improving their glycemic control. Automated telephone disease management (ATDM) systems can augment telephone care by providing frequent monitoring and health education to large patient panels while focusing clinicians� attention on individuals who need it most. Although this technology has shown some promise, it has not been rigorously evaluated, particularly in VA.

DETAILED DESCRIPTION:
Background:

Regular outpatient follow-up is important for all diabetes patients, with some needing frequent attention because their health is unstable, their treatment regimen is complex, or their social supports are inadequate. However, many patients live with access barriers that limit their use of outpatient services, fail to attend outpatient appointments, and experience worse outcomes than trials of aggressive management suggest is possible. Although labor-intensive, telephone care programs are one potential strategy for bringing diabetes management services into patients� homes and improving their glycemic control. Automated telephone disease management (ATDM) systems can augment telephone care by providing frequent monitoring and health education to large patient panels while focusing clinicians� attention on individuals who need it most. Although this technology has shown some promise, it has not been rigorously evaluated, particularly in VA.

Objectives:

This study evaluated Automated Telephone Disease Management (ATDM) calls with telephone nurse follow-up as a means of improving the quality of VA diabetes care. Specifically, we will determine whether this service improves patients' glucose control; improves other important outcomes such as their quality of life, satisfaction with care, and health service use; improves health behaviors such as self-monitoring of blood glucose, fat intake, and medication adherence; and has effects that vary across patient subgroups.

Methods:

Patients with diabetes mellitus using hypoglycemic medication were enrolled during outpatient visits to a university-affiliated VA health care system and randomized to usual care or bi-weekly ATDM assessment and self-care education calls with follow-up by a nurse educator. The intervention process was evaluated by examining patients� patterns of ATDM use and the reliability and validity of information they provided. Telephone surveys were used to measure intervention effects at 12-months on patients� self-care, symptoms, satisfaction with care, and perceived access barriers. The impact on VA utilization was evaluated using electronic utilization databases, and glycemic control was measured using laboratory tests. A total of 292 patients were randomized and 272 (93%) provided data at 12-months. Intervention patients completed ATDM assessments consistently throughout the observation period and the assessments identified groups of intervention patients with varying degrees of health risk at baseline. Compared to control patients, intervention patients at 12-months reported more frequent glucose self-monitoring, fewer access problems, and greater satisfaction with care (all p = 0.05). Intervention patients were more likely than controls to have been seen in podiatry clinics (53% versus 31%, p = 0.003) and diabetes specialty clinics (31% versus 17%, p = 0.03) during the study. The intervention did not influence mean endpoint HgA1c levels overall. However, among patients with baseline HgA1c = 8%, mean endpoint values among intervention and control patients were 8.7% and 9.2%, respectively (p = 0.05); intervention effects were even greater among patients with baseline HgA1c = 9%. Moreover, intervention patients at follow-up reported fewer symptoms of poor glycemic control than patients receiving usual care (3.6 versus 4.4, p = 0.03).

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

VA patients with diabetes taking hypoglycemic medications. Patients with serious mental disorders, no touch tone telephone, or a life expectancy of < 1 year were excluded.

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Study Completion 1999-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Piette, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, Michigan, United States

REFERENCES:
- [Result] Piette JD, McPhee SJ, Weinberger M, Mah CA, Kraemer FB. Use of automated telephone disease management calls in an ethnically diverse sample of low-income patients with diabetes. Diabetes Care. 1999 Aug;22(8):1302-9. doi: 10.2337/diacare.22.8.1302. PMID 10480775
- [Result] Piette JD. Patient education via automated calls: a study of English and Spanish speakers with diabetes. Am J Prev Med. 1999 Aug;17(2):138-41. doi: 10.1016/s0749-3797(99)00061-6. PMID 10490057
- [Result] Piette JD. Satisfaction with automated telephone disease management calls and its relationship to their use. Diabetes Educ. 2000 Nov-Dec;26(6):1003-10. doi: 10.1177/014572170002600613. PMID 11912804
- [Result] Piette JD. Perceived access problems among patients with diabetes in two public systems of care. J Gen Intern Med. 2000 Nov;15(11):797-804. doi: 10.1046/j.1525-1497.2000.91107.x. PMID 11119172
- [Result] Piette JD, Weinberger M, Kraemer FB, McPhee SJ. Impact of automated calls with nurse follow-up on diabetes treatment outcomes in a Department of Veterans Affairs Health Care System: a randomized controlled trial. Diabetes Care. 2001 Feb;24(2):202-8. doi: 10.2337/diacare.24.2.202. PMID 11213866
- [Result] Piette JD. Interactive voice response systems in the diagnosis and management of chronic disease. Am J Manag Care. 2000 Jul;6(7):817-27. PMID 11067378
- [Result] Piette JD. Satisfaction with care among patients with diabetes in two public health care systems. Med Care. 1999 Jun;37(6):538-46. doi: 10.1097/00005650-199906000-00003. PMID 10386566